CLINICAL TRIAL: NCT04576650
Title: Brain-Computer Interface Implant for Severe Communication Disability
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational device no longer available. No subjects enrolled.
Sponsor: Johns Hopkins University (Other)
Collaborators: UMC Utrecht (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00217299; U01DC016686 (NIH)
Record Dates: First submitted 2020-09-14; First posted 2020-10-06 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Locked-in Syndrome
MeSH Terms: conditions — Locked-In Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Summit system (Experimental): Implantation of Summit system, consisting of one or two Medtronic Activa(R) RC+S grids with wireless communication capabilities.
  Interventions: Device: Summit System

INTERVENTIONS:
Device: Summit System — Surgical implantation of the Summit system (consisting of one or two Medtronic Activa(R) RC+S grids with wireless communication capabilities) for Safety and efficacy testing of the Medtronic Summit System.

SUMMARY:
Locked-In Syndrome (LIS) is a devastating condition in which a person has lost the ability to communicate due to motor impairment, while being mentally intact. For people affected by this severe communication impairment, Brain-Computer Interfaces (BCI) may be the only solution that allows these people to start a conversation, ask questions, or request assistance (i.e. self-initiated communication). To-date, spelling was accomplished at a rate of 2-3 letters per minute with a predecessor device (the Medtronic Activa PC+S). To improve BCI performance, the current protocol will use the Medtronic Summit System, which offers a rechargeable battery and improved signal quality relative to Activa PC+S. Using signals from the motor hand/arm and/or motor mouth/face area, the investigators will investigate different avenues to improve the speed of communication using the Summit System. The primary objective is to evaluate the safety of the Summit System when used to chronically record subdural electrocorticographic (ECoG) signals in a BCI for use by patients with LIS in patients' homes. The secondary objective will be to evaluate the efficacy of the Summit System as a long-term source of ECoG signals for a BCI capable of allowing participants to control alternative and augmentative communication software in patients' homes.

DETAILED DESCRIPTION:
Locked-In Syndrome (LIS) is a devastating condition in which a person has lost the ability to communicate due to motor impairment, while being mentally intact. As a result, interaction with the environment is severely limited, and often can only be achieved in concert with a caregiver, who points at letters on a board one by one until the affected person blinks his or her eyes. For people affected by this severe communication impairment, Brain-Computer Interfaces (BCI) may be the only solution that allows these people to start a conversation, ask questions, or request assistance (i.e. self-initiated communication). A current study in the investigators' collaborator's lab at the University Medical Center Utrecht (UMCU, Utrecht, The Netherlands) aims to achieve communication in people with LIS, through a fully implantable BCI system, the Medtronic Inc. Activa PC+S. This is a research version of a deep brain stimulation device (Activa PC; FDA approved for treating Parkinson's disease and other disorders) that has been modified to allow electrophysiological recordings (+S for sensing). In the Utrecht Neuroprosthesis (UNP) study to date, spelling was accomplished at a rate of 2-3 letters per minute. To improve BCI performance, the current protocol will use the Medtronic Summit RC+S device (henceforth referred to as the Summit System), which offers a rechargeable battery and improved signal quality relative to Activa PC+S. Using signals from the motor hand/arm and/or motor mouth/face area, the investigators will investigate different avenues to improve the speed of communication. To achieve this, the investigators will use the Summit System under an investigational device exemption (IDE) and a Collaborative Research Agreement between Johns Hopkins University (JHU), UMCU, and Medtronic. The study has two main objectives. The primary objective is to evaluate the safety of the Summit System when used to chronically record subdural electrocorticographic (ECoG) signals in a BCI for use by patients with LIS in patients' homes. The secondary objective will be to evaluate the efficacy of the Summit System as a long-term source of ECoG signals for a BCI capable of allowing participants to control alternative and augmentative communication software in patients' homes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 22-75 years.
2. Clinical diagnosis of chronic Locked-In Syndrome (LIS) certified by an independent board-certified neurologist, defined here as impairments of voluntary motor control that are widespread and severe enough to prevent independent initiation and maintenance of communication, spoken or otherwise, without the assistance of a caregiver. Diagnosis of LIS requires exclusion of cognitive impairments as a cause for impaired communication (see Exclusion Criteria). For inclusion in this study, participants may have one of the following clinical variants of LIS:

   a. "Classic" Locked-In Syndrome, with the following signs documented on neurological examination i. Quadriplegia ii. Bulbar palsy iii. Anarthria iv. Partial or complete preservation of vertical eye movements and upper eyelid movements, or b. "Incomplete" Locked-In Syndrome, with the aforementioned signs of "Classic" LIS, documented on neurological examination, except that voluntary movements other than upper eyelid and vertical eye movement may be preserved, albeit still severe enough to prevent independent initiation and maintenance of communication, without the assistance of a caregiver. Preserved voluntary movements may include: i. Horizontal eye movements ii. Facial movements iii. Movements of the extremities not sufficient to reliably operate a joystick or mouse
3. Clinical diagnosis of, and confirmatory/exclusionary testing consistent with, one of the following irreversible or progressive neurological disorders as the cause for chronic Locked-In Syndrome, as defined above:

   a. Permanent lesion of corticospinal and corticobulbar tracts in the ventral pons (basis pontis) due to ischemic stroke, hemorrhage, or trauma, based on the following: i. Documented history of acute ischemic or hemorrhagic brainstem stroke or traumatic brainstem injury at onset of LIS ii. Ancillary testing including the following:

1. Brain MRI confirming a chronic lesion of the ventral pons, with no change on serial images at least 1 month apart, consistent with findings on neurological examination, involving at least 50% of the cross-sectional area on both sides of the basis pontis on at least one axial section 2. Absence of lesions on brain MRI that could contribute to communication impairment, including lesions of Broca's or Wernicke's areas, or sensorimotor cortex 3. EEG demonstrating posterior basic rhythm reactive to eye opening and closing iii. No clinical evidence of improving communication ability for at least 1 year prior to recruitment, confirming chronic LIS b. Diagnosis of Amyotrophic Lateral Sclerosis (ALS), certified by an independent board-certified neurologist with expertise in neuromuscular disorders, satisfying the following El Escorial World Federation of Neurology diagnostic criteria for probable, laboratory supported, or definite ALS: i. Signs of lower motor neuron (LMN) degeneration by neurological examination (weakness, atrophy, and fasciculations), electrophysiological (electromyographic findings of denervation), or neuropathological determination (muscle biopsy) in bulbar and at least two of three spinal regions (cervical, thoracic, lumbosacral), or in all three spinal regions ii. Signs of upper motor neuron (UMN) degeneration by clinical examination (spasticity, hyperreflexia, pseudobulbar affect, pathological reflexes) in bulbar and at least two of three spinal regions (cervical, thoracic, lumbosacral), or in all three spinal regions iii. Progressive spread of signs within a region or to other regions, together with the absence of electrophysiological or neuroimaging evidence of other disease processes that might explain clinical and electrophysiological signs of LMN and/or UMN degeneration (see below) iv. Confirmatory testing including:

1. Electrophysiological Studies

   1. Electromyographic findings of denervation (reduced recruitment, large motor unit action potentials, and fibrillation potentials) in clinically involved regions, including 3 of the following 4 muscle regions: bulbar, cervical, thoracic, and lumbosacral
   2. Nerve conduction studies confirming absence of demyelination as an explanation for aforementioned LMN signs
2. Neuroimaging, including brain and spine MRI, ruling out brain or spinal lesions (spinal cord or root compression) that could explain aforementioned LMN or UMN signs
3. Clinical laboratory examinations, determined by clinical judgment, to ascertain possible ALS-related syndromes v. History, physical, and laboratory examinations ruling out alternative diagnoses as cause of aforementioned clinical syndrome, including monoclonal gammopathy, autoimmune motor system degeneration, hyperthyroidism, hyperparathyroidism, paraneoplastic syndrome, infections of the central nervous system, toxic-metabolic disorders, or spinal cord injury due to trauma, electric shock, radiation therapy, vasculitis, ischemia, hemorrhage, or spondylotic myelopathy vi. No clinical evidence for improving communication ability for at least 6 months, confirming chronic LIS
4. Reliable means of communicating with caregiver(s) before entering the study, for example using vertical eye movements or eye blinking. Assessment of communication capabilities may be made by a physiatrist, a speech therapist, and/or an occupational therapist.
5. Residence within a reasonable driving distance from the JHU research team
6. Medically stable, including stable respiratory function, with or without artificial ventilation (see Section 12.2.3, Section 12.2.6, and Section 12.2.11).
7. Surgical clearance by the participant's primary healthcare provider, study physicians, and any necessary consultants
8. Stable psychosocial support system with caregiver(s) capable of monitoring the participant throughout the study. Caregivers must be willing and able to be present and provide routine care during all study activities except during hospitalization for device implantation.
9. Ability to understand and comply with study session instructions determined through the regular administration of simple study questionnaires.

Exclusion Criteria:

1. Strong and frequent muscle spasms not controlled by medication
2. Recent or remote history of brain tumor or tumor resection in any location
3. Cognitive impairments, according to neurological examination and neuropsychological testing, that contribute to impaired communication, or that could interfere with informed consent or participation in study activities
4. "Complete" Locked-In Syndrome without any voluntary movement, including vertical eye movements or blinking, without any reliable means of communicating with caregivers or others.
5. Known allergy to implanted materials
6. Contraindications to MRI prior to implantation (inability to lie flat in the scanner, MRI-incompatible metal objects in or attached to the body, claustrophobia)
7. Brain lesions that involve potential targets for implantation of BCI electrodes in sensorimotor cortical areas
8. No clearly identifiable targets for implantation of BCI electrodes after two pre-implantation functional magnetic resonance imaging (fMRI) localizer scans. Targets are identified as cortical areas of activation during attempted movements and/or speech.
9. Severe psychiatric illness that could interfere with informed consent or participation in study activities
10. Persistent suicidal ideation within the past 12 months or prior suicide attempt
11. Medical conditions contraindicating surgery or chronic device implantation
12. Treatment with immunosuppressive drugs
13. Chronic or acute medical condition that is anticipated to require surgery, radiotherapy, chemotherapy, immunosuppression, and/or MRI
14. Pregnant (confirmation through blood test), planning to become pregnant (sexually active without using effective birth control), or nursing an infant.
15. Visual impairment that would prevent use of computer monitor
16. Active cancer within the past year

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Safety of Summit System as assessed by the number of adverse events | Up to 52 weeks
  Record all adverse events on adverse events case report forms.
Safety of Summit System as assessed by change in neurological deficits | Immediately before device implantation, immediately after device implantation and 4-5 weeks after device implantation
  Pre- and post-surgical neurological/neurosurgical examinations to assess neurological deficits.
Safety of Summit System as assessed by the status of stimulation | Up to 52 weeks
  Verify that stimulation remains switched off (status is on or off).

SECONDARY OUTCOMES:
Efficacy of Summit System as assessed by change in letters spelled per minute | Weekly up to 52 weeks
  Letters spelled per minute while copying a 30 character sentence during weekly assessments.
Efficacy of Summit System as assessed by ability of participant to trigger the caregiver calling signal | Up to 52 weeks
  Ability to trigger the caregiver calling signal (yes or no) will be used in assessing the efficacy of the Summit System.
Change in Quality of Life as assessed by the ACSA | Every 12 weeks up to 52 weeks
  Change in responses to Anamnestic Comparative Self-Assessment (ACSA) every 12 weeks. This biographical +5 and -5 scale compares current quality of life to the participant's memories of the best period in their life and their worst period ever.
Frequency of use of Summit System per day | Up to 52 weeks
  Patterns of home use of the Summit system captured by logs of participants' use of the device

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Crone, MD, Principal Investigator — Professor of Neurology, Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States